CLINICAL TRIAL: NCT05169190
Title: Efficacy and Safety of Stellate Ganglion Block for Post-traumatic Stress Disorder in Veterans
Brief Title: Stellate Ganglion Block for PTSD
Acronym: SGB-PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Analydata, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-006-20F
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Veterans; Trauma Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a two-phase, three-arm (SGB vs Sham vs Wait List Control (WLC)), parallel-group (n=120 in each), triple-blind, prospective randomized controlled clinical trial (RCT). Phase I is 12-weeks and is the primary three-group RCT. Phase II is a 12-week open-label extension period where subjects in all groups are offered active SGB if eligible, defined as having PTSD scores > study inclusion criteria scores at the Phase I endpoints.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All assessments will be conducted by the Site Coordinator (SC) and clinical assessors at each time point blind to group allocation. The SGB assessor will conduct the Horner's syndrome evaluation after the procedure and will only share the results with data entry personnel. The primary data base in REDCap will show SID# only to keep the SC blinded while entering data. The minim program will assign each subject a Treatment ID number by site (e.g., TID# LB1S to LB20S for SGB at Long Beach site) and consecutive study ID numbers (e.g., SID# LB1 - LB90), which will be the only number on hard copies of documents in order to conceal allocation from all staff. The statisticians will be the only staff that will be able to link both SID and TID numbers to subject. The research pharmacy preparing the syringes will of course have both ID numbers and will label the syringes with only the SID#, keeping all personnel blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SGB (Active Comparator): SGB, the experimental procedure, is the injection of 7 cc of 0.5% ropivacaine plus 0.5 cc contrast anterior to the prevertebral fascia at the ventral aspect of the longus colli muscle, medial to Chassaignac's tubercle
  Interventions: Procedure: Stellate Ganglion Block
- Sham (Sham Comparator): Sham, the placebo control group, is the injection of 7 cc of normal saline plus 0.5 cc contrast anterior to the prevertebral fascia at the ventral aspect of the longus colli muscle, medial to Chassaignac's tubercle
  Interventions: Procedure: Sham Stellate Ganglion Block
- Wait-List Control (WLC) (No Intervention): WLC, a control for time, expectancy and safety, is all study procedures without going to the procedure room for injection

INTERVENTIONS:
Procedure: Stellate Ganglion Block — After procedure informed consent, the procedure will be done using an ultrasound guided technique with a high frequency (6 to 13 MHz) linear transducer and confirmation of placement by fluoroscopy at sites who do this in clinical practice. The subject will be prepped and draped and placed in supine position in a suite with continuous vital sign monitoring and advanced cardiac life support equipment and IV placement. Local anesthesia with 1% buffered lidocaine will be achieved. After visualization of Chassaignac's tubercle of C6 is identified along with the carotid artery, internal jugular vein and longus colli and capitus muscles, a 25-gauge echo-enhanced needle will be inserted to inject anesthetic over 2 minutes anterior to the prevertebral fascia at the ventral aspect of the longus colli muscle, medial to Chassaignac's tubercle. The needle will be withdrawn and the subject will be monitored for a minimum of 30 minutes.
  Other Names: SGB or Regional Block
  Arms: SGB
Procedure: Sham Stellate Ganglion Block — The Sham protocol is identical to the SGB protocol except "After needle tip confirmation and negative aspiration, normal saline (0.9%) + contrast (unlabeled to keep treater blinded) will be slowly injected over 2 minutes while closely monitoring the subject."
  Other Names: Sham SGB
  Arms: Sham

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a debilitating condition that affects about 15% of Veterans. Current treatments for Veterans with PTSD include medications and psychological therapies that help to process and desensitize to traumatic events. While effective for many, these treatments do not work for all patients, and many may refuse them. Stellate Ganglion Block (SGB), established to treat pain and other conditions, has shown promise for PTSD: early small studies show it may work fast and greatly reduce symptoms. However, data from larger studies are not clear about SGBs effects. A definitive trial is needed, especially for the Veteran population. This large, well-powered, randomized, sham-controlled trial of SGB for PTSD will assess the short-term efficacy of this intervention, the durability of the effects and the safety of the treatment. Additionally, this study will provide critically important information about biological effects of SGB and potential mechanisms of action. This timely study is critical to help VA clinicians better decide about the merits of SGB for PTSD.

DETAILED DESCRIPTION:
Stellate Ganglion Block (SGB) is a rapid-acting intervention that may directly target PTSD biology. Positive case-studies and preliminary results from the investigators' team suggest clinically robust and significant benefits for up to 6-months. Two randomized controlled trials, however, yielded conflicting results and had methodological limitations, making interpretation of results inconclusive. Neither trial evaluated durability beyond 8-weeks, safety, or biological mechanisms along with clinical outcomes. Veteran demand for SGB for PTSD is high, creating time-sensitive urgency for a more definitive study in VA. The investigators propose a 4-year, multi-site, two-phase, three-arm, (SGB-experimental condition, Sham-placebo control, Wait-List Control (WLC)-for time, expectancy and safety) parallel-group, triple-blind, prospective randomized controlled trial (RCT) of SGB for PTSD. The sample will include 360 treatment-seeking Veterans with chronic PTSD randomized 1:1:1 to the three arms using an adaptive randomization procedure. Phase I is a 12-week RCT with the primary aims of evaluating: a) within and between group differences in the change in PTSD symptom severity from pre- to 8-weeks post-intervention, b) durability of symptom reduction after SGB over 12 weeks, and c) safety (i.e., SGB will be as safe as Sham and WLC). Phase II is a 12-week open-label extension period where subjects in all groups are offered active SGB if eligible (PTSD scores > inclusion criteria scores at both primary Phase I endpoint of 8-weeks and durability endpoint of 12-weeks). Phase II is important because it allows evaluation of "enhanced dosing" (second SGB for those in the SGB arm), it allows all subjects to receive active intervention if they want, which also provides a larger sample of SGBs for exploratory pooled analyses, and it allows for analyses of durability over a longer time period for those in remission after Phase I. Another secondary aim is to test the hypothesis that SGB will be more biologically active than Sham or WLC by showing greater pre- to post-intervention reduction in highly PTSD-relevant fear-potentiated startle. The investigators will also explore clinical and biological phenotypic predictors of an SGB response (i.e., significant reduction in CAPS-5 scores). This superiority study is designed to expect and detect statistically and clinically important 30% PTSD symptom reduction from baseline to 8-week endpoint for SGB,15% reduction for Sham and 5% reduction for WLC in a sample with moderately severe PTSD (baseline score of 65+18). With these assumptions the investigators require a sample size of 262 subjects to test the primary hypothesis of clinical efficacy. The investigators will sample 360 subjects to account for 10% attrition, 5% missing data, a 5% failed-block rate and will oversample due to site variability. It is critical to ensure adequate power for this time-sensitive study. General linear mixed models (repeated multivariate analysis of variance (MANOVA)) will be used to evaluate the primary clinical hypothesized effects of intervention (SGB) on the clinical outcome of PTSD symptom severity (CAPS-5) over time (pre- to post-treatment to follow-up), controlling for baseline severity of symptoms and demographic characteristics (e.g., age, gender) in comparison with placebo control group (Sham) and WLC group with assumption of intent to treat while simultaneously adjusting for any significant covariates. Cohen's d within and between subjects will be calculated. Analyses will be performed on missing data due to loss-to-follow-up in order to determine if any potential bias exists once missing data are withdrawn. Details for analyses of the three primary aims are in the data analysis section of the Research Plan. The leadership team has extensive clinical and research experience with clinical trials, the use and adaptation of SGB for PTSD, and a national initiative to provide SGB to PTSD patients on a compassionate care basis. The proposed definitive study will guide rational use of SGB for PTSD in VA, will stimulate further research about dose, timing, biological mechanisms and clinical predictors of outcome, and will have established VA sites poised for further SGB research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Veterans of any military branch
* DSM-5 criteria for chronic PTSD on the Clinician Administered PTSD Scale (CAPS-5)
* at least moderate PTSD with a total CAPS-5 score of > 26
* having had at least one trial of an evidence-based treatment (EBT) for PTSD

Verification of an EBT trial will be by:

* subject report of engaging in the EBT (whether it be psycho- or pharmaco-therapy)
* CPRS or other medical record system (if outside VA) verification to determine that the dose and time (applies to both meds and therapy) was an adequate trial OR that they clearly did not finish the EBT due to clear aversion

  * They will be eligible if they did not finish the EBT due to aversion, but they must have had a trial and be fully informed during informed consent for this study of the available clinical treatment options
  * Eligible persons may have other symptoms that are commonly comorbid with PTSD (e.g., anxiety, moderate depression)
  * Severe primary depression will be an exclusion (see "Exclusion criteria" below)
  * This strategy will provide a feasible and generalizable sample
  * Women and minorities will be recruited

Exclusion Criteria:

* clear current and past six-months psychosis clearly not related to PSTD hypervigilance,
* substance dependence (clear evidence of tolerance and/or withdrawal) within the past 6 months
* thyroid disease and other contraindications to SGB (anatomic abnormalities of the anterior cervical spine; cardiac/pulmonary compromise; acute illness/infection; coagulopathy/bleeding disorder; allergic reactions/contraindications to local anesthetic or contrast dye, prior anterior neck surgery, anterior neck skin abnormalities (rash or eruptions))
* decisional incapacity (e.g., dementia, clear evidence of testing that signifies incapacity to consent), OR Montreal Cognitive Assessment score <18
* centrally acting medications that have a potential effect on biological expression
* pain levels requiring opiate medications
* known exposure to chemicals or physical trauma that cause permanent neuropsychiatric sequelae
* severe depression (Quick Inventory of Depression-SR16 (QIDS-SR16 score >18) that is deemed more clinically significant than PTSD (i.e., depression, cluster D PTSD, and minimal symptoms from cluster B, C, and E)
* high risk of acute suicidality
* a diagnosed and untreated moderate or severe sleep breathing disorder (SBD), OR a high risk of a SBD as indicated by snoring >50% of nights plus one of

  * any witnessed apnea
  * feeling non-refreshed in the morning >50% of mornings
  * daytime sleepiness indicated by falling asleep with routine tasks such as watching TV or reading
* clear treatment non-adherence indicated by stopping treatment or >3 missed appointments in the course of at least three PTSD EBTs
* past clear and chronic PTSD prior to military service
* current active psychotherapy for PTSD (they may suspend therapy if chosen by subject and therapist)
* pregnancy
* having had any prior SGB
* unstable dose(s) of medication for depression, anxiety, PTSD, or for sleep, or any other psychoactive medication for 8-weeks prior to intervention
* unwillingness to continue active medications at the same doses for the duration of the trial

  * a person who is on a stable medication dose for > 8 weeks who meets inclusion criteria and will continue these medications for the trial duration will not be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale-5 | 8 weeks after SGB, Sham, or WLC enrollment
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a structured diagnostic interview for PTSD. CAPS-5 items are rated with a single severity score, in contrast to previous versions of the CAPS which required separate frequency and intensity scores for each item that were either summed to create a symptom severity score or combined in various scoring rules to create a dichotomous (present/absent) symptom score. CAPS-5 has 20 symptom items, each rated from 0 (absent) to 4 (severe). There are 4 symptom clusters and DSM-5 diagnostic rule requires the presence of least one Criterion B symptom, one Criterion C symptom, two Criterion D symptoms, and two Criterion E symptoms in addition to other impairment criteria. A CAPS-5 cutoff score of >26 will be used for study inclusion.
Safety - Adverse Events and Side Effects from Treatment | 8 weeks after SGB, Sham, or WLC enrollment
  The Systematic Assessment for Treatment Emergent Events (SAFTEE) (Levine & Schooler, 1986) was developed at NIH and has been used in numerous clinical trials to track and compare adverse events and side-effects from pre- to post-intervention and between interventions. There is more than one version length. The investigators will use the 55-item version that has a baseline form and a "since last visit" form to comprehensively evaluate emergent symptoms in multiple body systems and compare pre- to post-intervention in a time X intervention approach.

SECONDARY OUTCOMES:
Peripheral Psychophysiology Startle Response | 8 weeks after SGB, Sham, or WLC enrollment
  Startle responses will be obtained from electromyographic (EMG) recordings during eyeblink muscle contractions elicited by a 108-dB burst of white noise that will be presented on each trial of the fear conditioning task. EMG startle eyeblink responses will be recorded using two 5mm Ag/AgCl electrodes placed over the orbicularis oculi muscle of the right eye. One electrode will be placed directly below the pupil in forward gaze while the other will be placed about 1 cm lateral to the first. Both electrodes will be placed as close to the eye as possible while still allowing the participant to close his or her eyes comfortably. Impedance between the two EMG electrodes will be measured and deemed acceptable if below 10 k .

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hollifield, MD, Principal Investigator — VA Long Beach Healthcare System, Long Beach, CA
Locations (6):
- United States (6):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollifield M, Brock C, Lim K, Holtzheimer P, Alkire M, Macedo F, Bovin MJ, Smith T, Romesser J, Messina M, Jovanovic T, Norrholm S, Krajec A. Efficacy and safety of the stellate ganglion block for posttraumatic stress disorder in veterans: Rationale for and methods of a multisite trial. Contemp Clin Trials. 2026 Jan;160:108180. doi: 10.1016/j.cct.2025.108180. Epub 2025 Dec 4. PMID 41352532

DOCUMENTS (1):
  • Informed Consent Form (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT05169190/ICF_000.pdf